CLINICAL TRIAL: NCT04578444
Title: Expanded Access Use of Zanidatamab for the Treatment of HER2-Positive Advanced Solid Tumor
Brief Title: An Expanded Access Treatment Protocol of Zanidatamab (ZW25) in Patients With HER2-Positive Advanced Biliary Tract Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ZWI-ZW25-EAP
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: HER2-Positive Advanced Biliary Tract Cancer
MeSH Terms: interventions — zanidatamab

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Zanidatamab — Administered intravenously
  Other Names: ZW25; ZIIHERA®

SUMMARY:
This is an intermediate-size Expanded Access Protocol (EAP) for use of zanidatamab (ZW25) in patients with human epidermal growth factor receptor 2 (HER2)-positive advanced biliary tract cancer (BTC) who are not eligible for other zanidatamab clinical trials, and who in the opinion of the treating oncologist, would potentially benefit from treatment with zanidatamab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HER2-positive locally advanced or metastatic biliary tract cancer that has progressed after receipt of available therapies known to confer clinical benefit.
* Adequate cardiac left ventricular function, as defined by left ventricular ejection fraction (LVEF) ≥ 50%
* Adequate organ function
* Ineligible to participate or has no access to an ongoing zanidatamab or other Zymeworks clinical study (e.g., ZW49 clinical study).
* Females of childbearing potential and non-sterile males must agree to practice highly effective methods of birth control for the duration of the study and for 12 months after the last dose of study drug. In addition, non-sterile males must avoid sperm donation for the duration of the study and for 12 months after the last dose of study drug.

Exclusion Criteria:

* Participating in other studies involving investigational drug(s) ≤ 3 weeks before the first dose of zanidatamab.
* Systemic anti-cancer therapy ≤ 3 weeks before the first dose of zanidatamab.
* Radiotherapy ≤ 2 weeks of the first dose of zanidatamab
* The following central nervous system (CNS) brain lesions are excluded from the study:

  * Untreated or unstable brain lesions requiring immediate local therapy or symptomatic CNS metastases.
  * Radiation treatment for CNS metastases within 4 weeks before the first dose of zanidatamab.
  * Known history of or ongoing leptomeningeal disease (LMD). If LMD has been reported radiographically, but is not suspected clinically by the investigator, the patient must be free of neurological symptoms of LMD.
  * The following CNS brain lesions are permitted:

    * Stable brain lesions are permitted if stable, as defined by patients who are off steroids and anticonvulsants and are neurologically stable with no evidence of radiographic progression for at least 4 weeks at the time of screening.
* Concurrent uncontrolled or active hepatobiliary disorders or untreated or ongoing complications after laparoscopic procedures or stent placement, including but not limited to active cholangitis, unresolved biliary obstruction, biloma or abscess. Any complications should be resolved within 2 weeks prior to the first dose of zanidatamab.
* Active hepatitis
* Infection with human immunodeficiency virus (HIV) with uncontrolled disease.
* Females who are breastfeeding or pregnant, and females and males planning a pregnancy.
* History of myocardial infarction or unstable angina within 6 months prior to enrollment, congestive heart failure (NYHA Class 3 or 4), or clinically significant cardiac disease
* QTc Fridericia (QTcF) > 470 ms assessed within 30 days of screening
* Acute or chronic uncontrolled pancreatitis or Child-Pugh Class C liver disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (17):
- United States (4):
  - NoCo Banner MD Anderson Cancer Center, Gilbert, Arizona
  - TOI Clinical Research, Cerritos, California
  - Salinas Valley Memorial Healthcare System, Salinas, California
  - Washington University School of Medicine, St Louis, Missouri
- France (4):
  - Jean Minjoz Hospital, Besançon
  - Hopital Timone Marseille, Marseille
  - Hopital Haut-Leveque - CHU Bordeaux, Pessac
  - Gustave Roussy Cancer Center, Villejuif
- Italy (3):
  - ICCRS Candiolo, Candiolo
  - Istituto Clinico Humanitas, Milan
  - Istituto Nazionale Tumori, Milan
- Spain (3):
  - Vall D'Hebron University Hospital, Barcelona
  - Fundacion Jimenez Diaz University Hospital - Autonomous University of Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (3):
  - The Princess Alexandra Hospital NHS Trust (Joanne Kwa, Pharmacist), Harlow
  - UCLH Cancer Institute (Meera Desai, Pharmacist), London
  - HCA Healthcare UK, London